CLINICAL TRIAL: NCT04526457
Title: Is Family Screening Improved by Genetic Testing of Familial Hypercholesterolemia
Acronym: IFIGhTFH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 820969
Record Dates: First submitted 2020-08-19; First posted 2020-08-25 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Hypercholesterolemia, Familial
Keywords: Familial Hypercholesterolemia; Genetics; Cascade screening
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Standard of Care; Genetic Testing

STUDY DESIGN:
Intervention Model Description: Probands were randomized 2:1 to genetic testing for FH plus lipid testing or lipid testing alone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Other): Participants with suspected FH (LDL-C greater than 220 mg/dL) or a previous clinical diagnosis of FH and randomized to standard of care with lipid testing only.
  Interventions: Other: Standard of Care
- Genetic Testing (Other): Participants with suspected FH (LDL-C greater than 220 mg/dL) or a previous clinical diagnosis of FH randomized to genetic testing
  Interventions: Other: Genetic Testing

INTERVENTIONS:
Other: Standard of Care — Randomized to standard of care with lipid testing only.
  Arms: Standard of Care
Other: Genetic Testing — Randomized to genetic testing.
  Arms: Genetic Testing

SUMMARY:
To test the hypothesis that in patients with a clinical diagnosis of familial hypercholesterolemia (FH), genetic testing and identification of a causative mutation might enhance the success of family-based cascade screening.

DETAILED DESCRIPTION:
To examine the impact of genetic testing on the efficiency of cascade screening for FH, patients with suspected FH or a clinical diagnosis of FH have been randomized to genetic testing or standard of care with lipid testing alone. After systematic encouragement of family enrollment, as a primary endpoint, the compared the number of probands with relatives enrolled in each group one year after results were returned to probands. The secondary endpoints examined include the number of relatives enrolled within 52 weeks of the genetic counseling call and the number of relatives diagnosed with FH through the study. Exploratory subgroup analyses were conducted stratifying the cohort by randomization/genetic test result. Further exploratory analyses compared probands' perceptions about high cholesterol diagnosis at baseline and at 20 weeks from enrollment

ELIGIBILITY:
Inclusion Criteria:

* For probands, inclusion criteria are as follows:

  1. LDL cholesterol > 220 mg/dL or a previous clinical diagnosis of FH
  2. Aged 18 years or older
  3. Ability to provide informed consent
  4. Willingness/ability to contact a minimum of 2 biological relatives about the study

Exclusion Criteria:

* For family members of probands, inclusion criteria are as follows:

  1. Willingness to participate in the study
  2. Age 10 or older
  3. Ability to give informed consent/assent

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Number of probands with relatives enrolled | 52 weeks after genetic/lipid testing results are returned to probands
  The primary outcome of this study was the number of probands with family members enrolled in the study within 52 weeks of results being returned to probands. Investigators compared the proportion of probands with a relative enrolled in the genetic testing group with the proportion of probands with a relative enrolled in the usual care group (lipid testing only). Relative enrolment was defined as the return of a test kit within the study time frame.

SECONDARY OUTCOMES:
The number of relatives enrolled in the study 52 weeks after results were returned to probands | 52 weeks after results are returned to probands
  The number of relatives enrolled in the study within 52 weeks of results being returned to probands. Investigators compared the number of relatives enrolled in the genetic testing group with the number of relatives enrolled in the usual care group (lipid testing only). Relative enrolment was defined as the return of a test kit within the study time frame.
The number of family members diagnosed with FH 52 weeks after results were returned to probands | 52 weeks after results are returned to probands
  The number of family members diagnosed with FH within 52 weeks of results being returned to probands. Investigators compared the number of enrolled relatives diagnosed with FH in the genetic testing group with the number of enrolled relatives diagnosed with FH in the usual care group (lipid testing only). This diagnosis had to be made through the study. The number of enrolled relatives diagnosed with FH in each group was expressed as the new case per index case ratio (relatives diagnosed with FH/total number of index case). Relative enrolment was defined as the return of a test kit within the study time frame. The diagnosis of FH was based on meeting either genetic or the Make Early Diagnosis To Prevent Early Deaths (MEDPED) clinical criteria

OTHER OUTCOMES:
Proband perceptions about their high cholesterol including its etiology, management and heritability at 20 weeks after enrollment compared to baseline | 20 weeks after enrollment
  Proband perceptions about their high cholesterol including its etiology, management and heritability were examined at baseline and 20 weeks after enrollment, using a questionnaire administered at these time points. Investigators examined proband agreement/disagreement with statements about the etiology of their high cholesterol, its management and heritability in these questionnaires. Using this approach, investigators were able to determine the proportion of probands that agreed/disagreed with these statements, and could compare how these proportions differed between the groups of interest at baseline/follow-up and how these changed from baseline to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Rader, MD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No
IRB approval to share IPD was not obtained for this protocol at the time of the initial protocol submission. If this should be required as part of the peer review process, or after publication of the study results and application will be submitted for a protocol amendment to fulfill this request

REFERENCES:
- [Background] Abul-Husn NS, Manickam K, Jones LK, Wright EA, Hartzel DN, Gonzaga-Jauregui C, O'Dushlaine C, Leader JB, Lester Kirchner H, Lindbuchler DM, Barr ML, Giovanni MA, Ritchie MD, Overton JD, Reid JG, Metpally RP, Wardeh AH, Borecki IB, Yancopoulos GD, Baras A, Shuldiner AR, Gottesman O, Ledbetter DH, Carey DJ, Dewey FE, Murray MF. Genetic identification of familial hypercholesterolemia within a single U.S. health care system. Science. 2016 Dec 23;354(6319):aaf7000. doi: 10.1126/science.aaf7000. PMID 28008010
- [Background] Benn M, Watts GF, Tybjaerg-Hansen A, Nordestgaard BG. Familial hypercholesterolemia in the danish general population: prevalence, coronary artery disease, and cholesterol-lowering medication. J Clin Endocrinol Metab. 2012 Nov;97(11):3956-64. doi: 10.1210/jc.2012-1563. Epub 2012 Aug 14. PMID 22893714
- [Background] Mortensen MB, Kulenovic I, Klausen IC, Falk E. Familial hypercholesterolemia among unselected contemporary patients presenting with first myocardial infarction: Prevalence, risk factor burden, and impact on age at presentation. J Clin Lipidol. 2016 Sep-Oct;10(5):1145-1152.e1. doi: 10.1016/j.jacl.2016.06.002. Epub 2016 Jun 14. PMID 27678431
- [Background] De Backer G, Besseling J, Chapman J, Hovingh GK, Kastelein JJ, Kotseva K, Ray K, Reiner Z, Wood D, De Bacquer D; EUROASPIRE Investigators. Prevalence and management of familial hypercholesterolaemia in coronary patients: An analysis of EUROASPIRE IV, a study of the European Society of Cardiology. Atherosclerosis. 2015 Jul;241(1):169-75. doi: 10.1016/j.atherosclerosis.2015.04.809. Epub 2015 Apr 30. PMID 25997074
- [Background] Wald DS, Bangash FA, Bestwick JP. Prevalence of DNA-confirmed familial hypercholesterolaemia in young patients with myocardial infarction. Eur J Intern Med. 2015 Mar;26(2):127-30. doi: 10.1016/j.ejim.2015.01.014. Epub 2015 Feb 11. PMID 25682442
- [Background] Pang J, Poulter EB, Bell DA, Bates TR, Jefferson VL, Hillis GS, Schultz CJ, Watts GF. Frequency of familial hypercholesterolemia in patients with early-onset coronary artery disease admitted to a coronary care unit. J Clin Lipidol. 2015 Sep-Oct;9(5):703-8. doi: 10.1016/j.jacl.2015.07.005. Epub 2015 Jul 18. PMID 26350818
- [Background] Nordestgaard BG, Chapman MJ, Humphries SE, Ginsberg HN, Masana L, Descamps OS, Wiklund O, Hegele RA, Raal FJ, Defesche JC, Wiegman A, Santos RD, Watts GF, Parhofer KG, Hovingh GK, Kovanen PT, Boileau C, Averna M, Boren J, Bruckert E, Catapano AL, Kuivenhoven JA, Pajukanta P, Ray K, Stalenhoef AF, Stroes E, Taskinen MR, Tybjaerg-Hansen A; European Atherosclerosis Society Consensus Panel. Familial hypercholesterolaemia is underdiagnosed and undertreated in the general population: guidance for clinicians to prevent coronary heart disease: consensus statement of the European Atherosclerosis Society. Eur Heart J. 2013 Dec;34(45):3478-90a. doi: 10.1093/eurheartj/eht273. Epub 2013 Aug 15. PMID 23956253
- [Background] Programme WHOHG. Familial hypercholesterolaemia (FH) : report of a second WHO consultation, Geneva, 4 September 1998. 1999:This report is dedicated to the memory of Professo.
- [Background] CDC. Genomic tests by levels of evidence. Centers for Disease Control Office of Public Health Genomics. http://www.cdc.gov/genomics/gtesting/file/print/tier.pdf. Published 2013. Accessed August 23, 2016.
- [Background] Knowles JW, Rader DJ, Khoury MJ. Cascade Screening for Familial Hypercholesterolemia and the Use of Genetic Testing. JAMA. 2017 Jul 25;318(4):381-382. doi: 10.1001/jama.2017.8543. No abstract available. PMID 28742895
- [Background] Sturm AC, Knowles JW, Gidding SS, Ahmad ZS, Ahmed CD, Ballantyne CM, Baum SJ, Bourbon M, Carrie A, Cuchel M, de Ferranti SD, Defesche JC, Freiberger T, Hershberger RE, Hovingh GK, Karayan L, Kastelein JJP, Kindt I, Lane SR, Leigh SE, Linton MF, Mata P, Neal WA, Nordestgaard BG, Santos RD, Harada-Shiba M, Sijbrands EJ, Stitziel NO, Yamashita S, Wilemon KA, Ledbetter DH, Rader DJ; Convened by the Familial Hypercholesterolemia Foundation. Clinical Genetic Testing for Familial Hypercholesterolemia: JACC Scientific Expert Panel. J Am Coll Cardiol. 2018 Aug 7;72(6):662-680. doi: 10.1016/j.jacc.2018.05.044. PMID 30071997
- [Background] Umans-Eckenhausen MA, Defesche JC, Sijbrands EJ, Scheerder RL, Kastelein JJ. Review of first 5 years of screening for familial hypercholesterolaemia in the Netherlands. Lancet. 2001 Jan 20;357(9251):165-8. doi: 10.1016/S0140-6736(00)03587-X. PMID 11213091
- [Background] Leren TP, Finborud TH, Manshaus TE, Ose L, Berge KE. Diagnosis of familial hypercholesterolemia in general practice using clinical diagnostic criteria or genetic testing as part of cascade genetic screening. Community Genet. 2008;11(1):26-35. doi: 10.1159/000111637. Epub 2008 Jan 15. PMID 18196915
- [Background] Nherera L, Marks D, Minhas R, Thorogood M, Humphries SE. Probabilistic cost-effectiveness analysis of cascade screening for familial hypercholesterolaemia using alternative diagnostic and identification strategies. Heart. 2011 Jul;97(14):1175-81. doi: 10.1136/hrt.2010.213975. PMID 21685482
- [Background] deGoma EM, Ahmad ZS, O'Brien EC, Kindt I, Shrader P, Newman CB, Pokharel Y, Baum SJ, Hemphill LC, Hudgins LC, Ahmed CD, Gidding SS, Duffy D, Neal W, Wilemon K, Roe MT, Rader DJ, Ballantyne CM, Linton MF, Duell PB, Shapiro MD, Moriarty PM, Knowles JW. Treatment Gaps in Adults With Heterozygous Familial Hypercholesterolemia in the United States: Data From the CASCADE-FH Registry. Circ Cardiovasc Genet. 2016 Jun;9(3):240-9. doi: 10.1161/CIRCGENETICS.116.001381. Epub 2016 Mar 24. PMID 27013694
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2889-934. doi: 10.1016/j.jacc.2013.11.002. Epub 2013 Nov 12. No abstract available. PMID 24239923
- [Derived] Ajufo E, deGoma EM, Raper A, Yu KD, Cuchel M, Rader DJ. A randomized controlled trial of genetic testing and cascade screening in familial hypercholesterolemia. Genet Med. 2021 Sep;23(9):1697-1704. doi: 10.1038/s41436-021-01192-z. Epub 2021 May 26. PMID 34040191